CLINICAL TRIAL: NCT01882296
Title: A Block-randomized, Open-Label, Multiple Oral Dosing, Phase I Study to Explore Comparability of the Pharmacodynamics Between S-pantoprazole 10, 20, 40mg and Pantoprazole 20, 40mg in Healthy Male Subjects
Brief Title: Investigate a Pharmacodynamics Between S-pantoprazole 10, 20, 40mg and Pantoprazole 20, 40mg in Healthy Male Subjects
Acronym: AGSPT_PD
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ahn-Gook Pharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AGSPT_PD
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-05

CONDITIONS: Healthy Male Subjects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- AGSPT_10 (Experimental): tablet, 10mg, QD, 7days
  Interventions: Drug: AGSPT_10
- AGSPT_20 (Experimental): tablet, 20mg, QD, 7days
  Interventions: Drug: AGSPT_20
- AGSPT_40 (Experimental): tablet, 20mg x 2, QD, 7days
  Interventions: Drug: AGSPT_40
- Pantoprazole_20 (Active Comparator): tablet, 20mg, QD, 7days
  Interventions: Drug: Pantoprazole_20
- Pantoprazole_40 (Active Comparator): tablet, 40mg, QD, 7days
  Interventions: Drug: Pantoprazole_40

INTERVENTIONS:
Drug: AGSPT_10 — AGSPT 10mg for 7days administration
  Arms: AGSPT_10
Drug: AGSPT_20 — AGSPT 20mg for 7days administration
  Arms: AGSPT_20
Drug: AGSPT_40 — AGSPT 20mg x 2tablet for 7days administration
  Arms: AGSPT_40
Drug: Pantoprazole_20 — Pantoprazole 20mg for 7days administration
  Arms: Pantoprazole_20
Drug: Pantoprazole_40 — Pantoprazole 40mg for 7days administration
  Arms: Pantoprazole_40

SUMMARY:
Primary object: Evaluate Pharmacodynamic property and safety administered S-pantoprazole 10, 20, 40mg and Pantoprazole 20, 40mg in healthy male subjects

Secondary object : Evaluate Dose-response of S-pantoprazole and pantoprazole and compare each dose-response

ELIGIBILITY:
Inclusion Criteria:

* Adult healthy males 20 to 45 years at screening
* BMI : 19kg/m2 ~ 26 kg/m2
* Blood Pressure : "140 mmHg ≥ sitting SBP ≥ 90 mmHg, 95 mmHg ≥ sitting DBP ≥ 50 mmHg"

Exclusion Criteria:

* Have history of significant hepatic, renal gastrointestinal, pulmonary, musculoskeletal, endocrine, neuropsychiatric, hematologic, cardiovascular diseases
* Have a gastrointestinal disease(ex : Crohn's disease, gastrointestinal ulcer) or surgery (except for Appendectomy, hernia repair) affected the absorption of medications
* Have history of GERD, Gastric ulcer, Duodenal ulcer and H.pylori positive
* Hypersensitivity reactions to drugs of clinically significant hypersensitivity reactions in the history of benzimidazole (ex: pantoprazole, NSAID, antibiotic)
* Have a history of drug abuse
* unusual diet affected the absorption, distribution, metabolism, excretion of medications
* Subject who treated with any investigational drugs within 90 days before the administration of investigational drug
* Subject who takes inhibitors and inducers of drug metabolizing enzyme (Barbiturates etc.) within 30days
* Previously donate whole blood within 60 days or component blood within 30 days or transfusion within 30 days
* Subject who have taken habitually caffeine (caffeine > 5 units/day)
* Subject who have drunken habitually (alcohol > 21 units/week, 1 unit = pure alcohol 10ml)or who are unable to quit drinking during this study or smoker
* Subjects deemed ineligible by investigator based on other reasons

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Primary Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
24h pH | 24 hours

SECONDARY OUTCOMES:
%Time pH>6 | 24 hours
  (Time(hour) percent when pH >6) / 24(hours)
% inhibition time gastric pH≤4 | 24 hours
  100-(percent time pH >4)